CLINICAL TRIAL: NCT02255851
Title: Histopathology of Embolic Debris Captured During Transcatheter Aortic Valve Replacement
Brief Title: Sentinel(TM) Post-Market Registry
Status: Completed | Type: Observational
Sponsor: Claret Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CP10879
Record Dates: First submitted 2014-09-25; First posted 2014-10-03 (Estimated); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Transcatheter Aortic Valve Replacement; Severe Symptomatic Calcified Native Aortic Valve Stenosis
Keywords: selected for TAVR by heart team consensus; treated with CE-Marked TAVR devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Capture and histopathology analysis of embolic debris. (Thrombus, valve tissue, amorphous calcium, etc.)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment Group: TAVR + SENTINEL (Cerebral Protection System)
  Interventions: Device: SENTINEL (Cerebral Protection System)

INTERVENTIONS:
Device: SENTINEL (Cerebral Protection System)

SUMMARY:
The SENTINEL Post-Market Registry is a prospective, multi-center, registry using the CE-Marked Sentinel System in subjects with severe symptomatic calcified native aortic valve stenosis indicated for TAVR.

Subjects enrolled in the registry will undergo TAVR + Sentinel. Basic demographic information and detailed procedural data will be captured and documented in a registry case report form.

All Sentinel filters will be sent for histopathology at an independent core-lab.

ELIGIBILITY:
Inclusion Criteria:

1. Approved indications for commercially available CE-Marked TAVR devices.
2. Compatible left common carotid artery (6.5 - 10 mm) and brachiocephalic artery (9 - 15 mm) diameters without significant stenosis (> 70%).
3. The subject or the subject's legal representative has been informed of the nature of the registry, agrees to its provisions and has provided written informed consent as approved by the Ethics Committee of the respective site.

Exclusion Criteria:

1. Vasculature in the right extremity precluding 6Fr sheath radial/brachial access
2. Inadequate circulation to the right extremity as evidenced by signs of artery occlusion or absence of radial or brachial pulse
3. Hemodialysis shunt, graft, or arterio-venous fistula involving the upper extremity vasculature
4. Patients in whom anti-platelet and/or anticoagulant therapy is contraindicated, or who will refuse transfusion
5. Excessive tortuosity in the right radial/brachial/subclavian artery preventing Sentinel device access and insertion
6. Patient whose brachiocephalic or left carotid artery reveals significant stenosis, ectasia, dissection, or aneurysm at the ostium or within 3 cm of the ostium
7. Currently participating in an investigational drug or investigational (non CE-mark) device study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The registry population comprises subjects with severe symptomatic calcified native aortic valve stenosis who are selected for TAVR by heart team consensus and treated with CE-Marked TAVR devices.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Primary Observational Endpoint | Post-Procedure (day 1)
  Capture rate, debris volume and histopathology analysis at day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Naber, MD, Principal Investigator — Elisabeth-Krankenhaus Essen GmbH, Essen, Germany